CLINICAL TRIAL: NCT05559879
Title: A Phase Ib/II Single Arm Study of Cabozantinib Plus Dostarlimab in Women With Recurrent Gynecologic Carcinosarcoma
Brief Title: Cabozantinib and Dostarlimab in Recurrent Gynecologic Carcinosarcoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Michael Toboni, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300008749 (UAB21111); 000547299 (Other: GSK and Exelixis)
Record Dates: First submitted 2022-08-29; First posted 2022-09-29 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Gynecologic Cancer; Carcinoma; Uterine Cancer; Endometrial Cancer
Keywords: Gynecologic Cancer; Carcinoma; Uterine Cancer; Endometrial Cancer
MeSH Terms: conditions — Carcinoma; Uterine Neoplasms; Endometrial Neoplasms | interventions — VMBP protocol; dostarlimab

STUDY DESIGN:
Intervention Model Description: This is a phase Ib/II, single-arm, combination therapy of the safety and efficacy of therapy involving a tyrosine kinase inhibitor along with immunotherapy in the setting of recurrent carcinosarcoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cabo + Dostarlimab (Experimental): Cabozantinib 40 mg by mouth every day + Dostarlimab 500 mg intravenous every 3 weeks followed by maintenance therapy: Cabozantinib 40 mg by mouth every day + Dostarlimab 1000 mg intravenous every 6 weeks
  Interventions: Drug: Cabo + Dostarlimab

INTERVENTIONS:
Drug: Cabo + Dostarlimab — Combination of standard dose of cabozantinib and 500 mg dostarlimab for first 4 cycles followed by standard dose of cabozantinib and 1000 mg of dostarlimab until 2 years of treatment

SUMMARY:
Immunotherapy has gained a significant amount of attention recently, but its efficacy as a single agent in gynecological cancers has been disappointing. Pre-clinical evidence supports the combination of using Vascular Endothelial Growth Factors (VEGF) inhibitors with immunotherapy. VEGF inhibitors suppress the activation of tumor-associated macrophages (TAMs) and VEGF has been shown to affect the functional maturation of dendritic cells; therefore, VEGF inhibitors could improve the function of antigen presentation. In this study, Cabozantinib (VEGF inhibitor) and Dostarlimab (immunotherapeutic drug) will be admnistered as a combination to patients with recurrent gynecologic carcinosarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of carcinosarcoma (independent of organ of gynecologic origin)
2. Received at least one prior chemotherapy regimen for their cancer
3. Must have measurable or evaluable lesion defined by iRECIST
4. Recovery to baseline or ≤ Grade 1 CTCAE v5.0 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy
5. ECOG Performance Status of 0-2
6. Age ≥ 18 years
7. Adequate organ and marrow function, based upon meeting all of the following laboratory criteria within 14 days before first dose of study treatment:

   1. Absolute neutrophil count (ANC) ≥ 1500/mm3 (≥ 1.5 GI/L) without granulocyte colony-stimulating factor support.
   2. White blood cell count ≥ 2500/mm3 (≥ 2.5 GI/L).
   3. Platelets ≥ 100,000/mm3 (≥ 100 GI/L) without transfusion.
   4. Hemoglobin ≥ 9 g/dL (≥ 90 g/L).
   5. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 x upper limit of normal (ULN). ALP ≤ 5 x ULN with documented bone metastases.
   6. Total bilirubin ≤ 1.5 x ULN (for patients with Gilbert's disease ≤ 3 x ULN).
   7. Serum albumin ≥ 2.8 g/dl.
   8. Serum creatinine ≤ 2.0 x ULN or calculated creatinine clearance ≥ 30 mL/min (≥ 0.5 mL/sec) using the Cockcroft-Gault equation:

   [(140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)] × 0.85 i. Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol).
8. Capable of understanding and complying with the protocol requirements and must have signed the informed consent document.
9. Women of childbearing potential (WOCBP) ie. sexually active fertile patients and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 5 months after the last dose of study treatment.
10. Females should not breastfeed while receiving treatment on trial.
11. Female patients of childbearing potential must not be pregnant at screening. Females of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e., females who have had any evidence of menses in the past 12 months, with the exception of those who had a prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression, or other reasons.

Exclusion Criteria:

1. Prior treatment with cabozantinib.
2. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks or 5 half-lives (whichever is longer) before first dose of study treatment.
3. Receipt of any type of cytotoxic, biologic, or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment.
4. Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before the first dose of study treatment. Patients with clinically relevant ongoing complications from prior radiation therapy are not eligible.
5. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment. Eligible patients must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment.
6. Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixabin, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

   1. Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
   2. Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
7. The patient has prothrombin time (PT)/INR or partial thromboplastin time (PTT) test ≥ 1.3 X the laboratory ULN within 7 days before the first dose of study treatment.
8. The patient has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   a. Cardiovascular disorders: i. Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.

   ii. Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.

   iii. Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose.

   b. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation: i. The patient has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.

   ii. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose.

   Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose.

   c. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose.

   d. Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.

   e. Lesions invading or encasing any major blood vessels. f. Other clinically significant disorders that would preclude safe study participation.

   i. Serious non-healing wound/ulcer/bone fracture ii. Uncompensated/symptomatic hypothyroidism (i.e. inadequately treated hypothyroidism) iii. Moderate to severe hepatic impairment (Child-Pugh B or C)
9. Major surgery (e.g., laparoscopic nephrectomy, GI surgery, removal or biopsy of brain metastasis) within 2 weeks before first dose of study treatment. Minor surgeries within 10 days before first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
10. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 28 days before first dose of study treatment [add reference for Fridericia formula].

    Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.
11. Inability to swallow tablets.
12. Previously identified allergy or hypersensitivity to components of the study treatment formulations.
13. Diagnosis of another malignancy within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy.
14. Patients with concurrent cytotoxic chemotherapy or radiation therapy are excluded.
15. Patients with a serious chronic or acute illness, such as cardiac disease (NYHA class III or IV), hepatic disease, or other illness considered by the Principal Investigator as unwarranted high risk for investigational drug treatment.
16. Patients with a medical or psychological impediment to probable compliance with the protocol should be excluded.
17. Presence of a known active acute or chronic infection including: a urinary tract infection, HIV or viral hepatitis; however, it is acceptable to treat an acute infection and then re-screen or re-evaluate eligibility.
18. Administration of a live, attenuated vaccine within 30 days prior to first dose of study treatment
19. Other clinically significant disorders:

    1. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
    2. Active, known, or suspected autoimmune disease (exceptions: type 1 diabetes mellitus, hypothyroidism, skin disorders, conditions not expected to recur in the absence of an external trigger)
    3. Malabsorption syndrome
    4. Requirement for hemodialysis or peritoneal dialysis
    5. History of solid organ or allogenic stem cell transplant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 37 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival at 6 months | 6 months
  To estimate the proportion of patients with recurrent carcinosarcoma-who survive progression-free for at least 6 months from the start of treatment-treated with cabozantinib + dostarlimab in the second line setting and beyond (per imaging Response Evaluation Criteria in Solid Tumours).

CONTACTS AND LOCATIONS:
Locations (1):
- O'Neal Comprehensive Cancer Center at UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided